CLINICAL TRIAL: NCT04556630
Title: Evaluation of the Experience of Lock Down Related to the Covid-19 Epidemic and Its Impact on the Project of Parenthood of the Couples Followed in Assisted Reproduction
Brief Title: Experience of Lock Down Related to the Covid-19 Epidemic and Its Impact on the Project of Parenthood
Acronym: CONFIN-AMP
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_65; 2020-A01810-39 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-09-18; First posted 2020-09-21 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Assisted Reproduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational, descriptive, cross-sectional, monocentric study, This Study is proposed to all couples followed in Assisted Reproduction and CECOS Nord for whom the protocols were stopped when they entered into confinement related to the Covid-19 epidemic on 13 March 2020.

ELIGIBILITY:
Inclusion Criteria:

* couples followed up in Assisted Reproduction and CECOS Nord
* the cessation of assistance reproduction protocols related to the Covid-19 outbreak on March 13, 2020.
* acceptance of teleconsultation

Exclusion Criteria:

* Individuals refusing to participate in the study during the teleconsultation with the referring practitioner.

I- ndividuals who do not respond to the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: couples followed up in Assisted Reproduction and CECOS Nord
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Level of anxiety and/or depression of MPA patients (male and female couples) by Hospital Anxiety and Depression Scale (HAD) score. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bérengère DUCROCQ, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Calmette Chu Lille, Lille, France